CLINICAL TRIAL: NCT02556034
Title: Assessment of Tender & Swollen Joints Count Score Performed by a Rheumatologist And Rheumatology Nurses in Patients With Rheumatoid Arthritis (RA) and Psoriatic Arthritis (PsA)
Brief Title: Assessment of Tender & Swollen Joints Count Score Performed by a Rheumatologist And Rheumatology Nurses in Patients With RA and PsA.
Acronym: APRAN
Status: Completed | Type: Observational
Sponsor: Isabelle Fortin (Other)
Collaborators: Janssen Inc. (Industry)
Responsible Party: Sponsor-Investigator, Isabelle Fortin, Rheumatologist, Centre de Rhumatologie de l'Est du Québec
Organization: Centre de Rhumatologie de l'Est du Québec (Other)
Other Study IDs: CNTO148ART4009
Record Dates: First submitted 2015-09-15; First posted 2015-09-22 (Estimated); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Rheumatoid Arthritis; Psoriatic Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis, Psoriatic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Disease evaluation: Rheumatoid arthritis evaluations.
  Interventions: Other: Disease evaluation.

INTERVENTIONS:
Other: Disease evaluation. — Patients will complete a self-evaluation of 28 joint counts for swelling and tenderness and assess their disease activity on a Visual Analog Scale. A 28 joint count and VAS will then be assessed by a nurse and by a rheumatologist. The same rheumatologist will examine all patients and two nurses will each randomly assess half the total enrolled patients. The nurse will be blinded to the patient's joint count and VAS, and similarly, the rheumatologist will be blinded to both the patient and nurse's assessments.

SUMMARY:
This study will establish a comparison in follow-up care of 100 patients between Health Care Practitioners, more specifically the rheumatologist and a trained nurse. The study objective is to show consistency of evaluation between two different health care professionals, a physician and a nurse.

DETAILED DESCRIPTION:
This study involves one site in Canada. Patients will complete a self-evaluation of 28 joint counts for swelling (SJC) and tenderness (TJC) and assess their disease activity on a Visual Analog Scale (VAS). A 28 joint count and VAS will then be assessed by a nurse and by a rheumatologist. Clinical Disease Activity Index (CDAI) and Disease Activity Severity 28 - C Reactive protein (DAS28-CRP) will be calculated from each data set.

The same rheumatologist will examine all patients and two nurses will each randomly assess half the total enrolled patients. The nurse will be blinded to the patient's joint count and VAS, and similarly, the rheumatologist will be blinded to both the patient and nurse's assessments. The setting includes 2 nurses with different educational background: one technician and one bachelor.

The training provided to the nurses in this study allows them to master the basis of the physical exam, joint count and history of the rheumatoid patient as well as to learn the pertinent laboratory parameters. It is a 14-hour course in which the patient is examined through observation, palpation, assessment of mobility and stability and specific movement. Diagnostic tools such as the Simplified Disease Activity Index (SDAI), Health Assessment Questionnaire Disability Index (HAQ), CDAI and DAS-28 are included in the patient evaluation.

Each enrolled patient will receive a 5-minute training in joint assessment by the nurse. The use of the mannequin for joint assessment of swelling and tenderness will be reviewed. Objective signs of disease such as swelling, redness and heat will be explained as well as the difference between inflammation and bony swelling, the latter being indicative of osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥18 years of age.
2. Has at least one of the following diagnosis at screening

   * Subject has a diagnosis of RA as defined by the 1987- revised American College of Rheumatology (ACR)- classification criteria for RA and has disease duration of more than 6 months.
   * Subject must have a diagnosis of active PsA by Classification Criteria for Psoriatic Arthritis (CASPAR) and has disease duration of more than 6 months.
3. The subject must be able to provide written informed consent and to complete the study questionnaires.

Exclusion Criteria:

* Subject with DIP involvement in PsA
* Subject with predominant axial symptoms (spondyloarthropathy)
* Subject with fibromyalgia
* Subject involved in a concomitant study
* Subject currently takes ≥10 mg cortisone daily
* Subject has taken opioid analgesics within 12 hours of joint count assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The target population will be subjects with active Rheumatoid Arthritis or Psoriatic Arthritis.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2015-09; Primary Completion 2018-11-16 (Actual); Study Completion 2018-11-16 (Actual)

PRIMARY OUTCOMES:
Accuracy of the nurse CDAI result compared to the rheumatologist CDAI result. | 6 months
  To validate the accuracy of assessment of RA and PsA disease activity by a nurse trained in joint examination using the CDAI as compared to a rheumatologist's same assessment. The level of agreement between evaluators will be investigated using Cohen's Kappa, a statistic tool useful to the measurement of inter-rater agreement for qualitative traits.
Accuracy of the nurse DAS-28 result compared to the rheumatologist DAS-28 result. | 6 months
  To validate the accuracy of assessment of RA and PsA disease activity by a nurse trained in joint examination using the DAS-28 as compared to a rheumatologist's same assessment. The level of agreement between evaluators will be investigated using Cohen's Kappa, a statistic tool useful to the measurement of inter-rater agreement for qualitative traits.

SECONDARY OUTCOMES:
Comparison of TJC results between 3 raters. | 6 months
  The TJC results from the patient self-assessment, nurse assessment and physician assessment are compared.
Comparison of SJC results between 3 raters. | 6 months
  The SJC results from the patient self-assessment, nurse assessment and physician assessment are compared.
Comparison of VAS results between 3 raters. | 6 months
  The VAS results from the patient self-assessment, nurse assessment and physician assessment are compared.
Comparison of time taken by 3 raters to perform disease assessments. | 6 months
  To compare the time taken by the rheumatologist, nurse and patient to complete each part of the joint count assessment and the VAS. An ANOVA will be used to verify if a significant difference is present in the assessment time between the different raters.

CONTACTS AND LOCATIONS:
Overall Officials: NABIL CHAKER, BIOLOGIST, Study Director — CENTRE DE RHUMATOLOGIE DE L'EST DU QUEBEC; ISABELLE FORTIN, MD, Principal Investigator — CENTRE DE RHUMATOLOGIE DE L'EST DU QUEBEC; FRÉDÉRIC BANVILLE, Ph.D, Principal Investigator — Université de Montréal
Locations (1):
- Centre de Rhumatologie de L'Est Du Quebec, Rimouski, Quebec, Canada

REFERENCES:
- [Result] Smolen JS, Aletaha D, Bijlsma JW, Breedveld FC, Boumpas D, Burmester G, Combe B, Cutolo M, de Wit M, Dougados M, Emery P, Gibofsky A, Gomez-Reino JJ, Haraoui B, Kalden J, Keystone EC, Kvien TK, McInnes I, Martin-Mola E, Montecucco C, Schoels M, van der Heijde D; T2T Expert Committee. Treating rheumatoid arthritis to target: recommendations of an international task force. Ann Rheum Dis. 2010 Apr;69(4):631-7. doi: 10.1136/ard.2009.123919. Epub 2010 Mar 9. PMID 20215140
- [Result] Atar D, Birkeland KI, Uhlig T. 'Treat to target': moving targets from hypertension, hyperlipidaemia and diabetes to rheumatoid arthritis. Ann Rheum Dis. 2010 Apr;69(4):629-30. doi: 10.1136/ard.2010.128462. No abstract available. PMID 20237122
- [Result] Anderson J, Caplan L, Yazdany J, Robbins ML, Neogi T, Michaud K, Saag KG, O'Dell JR, Kazi S. Rheumatoid arthritis disease activity measures: American College of Rheumatology recommendations for use in clinical practice. Arthritis Care Res (Hoboken). 2012 May;64(5):640-7. doi: 10.1002/acr.21649. PMID 22473918
- [Result] Scott IC, Scott DL. Joint counts in inflammatory arthritis. Clin Exp Rheumatol. 2014 Sep-Oct;32(5 Suppl 85):S-7-12. Epub 2014 Oct 30. PMID 25365082
- [Result] Radner H, Grisar J, Smolen JS, Stamm T, Aletaha D. Value of self-performed joint counts in rheumatoid arthritis patients near remission. Arthritis Res Ther. 2012 Mar 14;14(2):R61. doi: 10.1186/ar3777. PMID 22417647
- [Result] Cheung PP, Ruyssen-Witrand A, Gossec L, Paternotte S, Le Bourlout C, Mazieres M, Dougados M. Reliability of patient self-evaluation of swollen and tender joints in rheumatoid arthritis: A comparison study with ultrasonography, physician, and nurse assessments. Arthritis Care Res (Hoboken). 2010 Aug;62(8):1112-9. doi: 10.1002/acr.20178. PMID 20235213
- [Result] Tillett W, Shaddick G, Korendowych E, de Vries CS, McHugh N. Joint count reliability in psoriatic arthritis observational trials--an unreported problem. Rheumatology (Oxford). 2012 Jul;51(7):1333-4. doi: 10.1093/rheumatology/kes095. Epub 2012 May 4. No abstract available. PMID 22562935
- [Result] Janta I, Naredo E, Martinez-Estupinan L, Nieto JC, De la Torre I, Valor L, Estopinan L, Bello N, Hinojosa M, Gonzalez CM, Lopez-Longo J, Monteagudo I, Montoro M, Carreno L. Patient self-assessment and physician's assessment of rheumatoid arthritis activity: which is more realistic in remission status? A comparison with ultrasonography. Rheumatology (Oxford). 2013 Dec;52(12):2243-50. doi: 10.1093/rheumatology/ket297. Epub 2013 Sep 17. PMID 24046468
- [Result] Barton JL, Criswell LA, Kaiser R, Chen YH, Schillinger D. Systematic review and metaanalysis of patient self-report versus trained assessor joint counts in rheumatoid arthritis. J Rheumatol. 2009 Dec;36(12):2635-41. doi: 10.3899/jrheum.090569. Epub 2009 Nov 16. PMID 19918045
- [Result] Levy G, Cheetham C, Cheatwood A, Burchette R. Validation of patient-reported joint counts in rheumatoid arthritis and the role of training. J Rheumatol. 2007 Jun;34(6):1261-5. Epub 2007 Apr 15. PMID 17444590
- [Result] Cheung PP, Dougados M, Andre V, Balandraud N, Chales G, Chary-Valckenaere I, Dernis E, Gill G, Gilson M, Guis S, Mouterde G, Pavy S, Pouyol F, Marhadour T, Richette P, Ruyssen-Witrand A, Soubrier M, Nguyen M, Gossec L. The learning curve of nurses for the assessment of swollen and tender joints in rheumatoid arthritis. Joint Bone Spine. 2014 Mar;81(2):154-9. doi: 10.1016/j.jbspin.2013.06.006. Epub 2013 Aug 6. PMID 23928236
- [Result] Farragher TM, Lunt M, Plant D, Bunn DK, Barton A, Symmons DP. Benefit of early treatment in inflammatory polyarthritis patients with anti-cyclic citrullinated peptide antibodies versus those without antibodies. Arthritis Care Res (Hoboken). 2010 May;62(5):664-75. doi: 10.1002/acr.20207. PMID 20461787
- [Result] Pincus T, Segurado OG. Most visits of most patients with rheumatoid arthritis to most rheumatologists do not include a formal quantitative joint count. Ann Rheum Dis. 2006 Jun;65(6):820-2. doi: 10.1136/ard.2005.044230. Epub 2005 Nov 16. PMID 16291813
- [Result] Cheung PP, Gossec L, Mak A, March L. Reliability of joint count assessment in rheumatoid arthritis: a systematic literature review. Semin Arthritis Rheum. 2014 Jun;43(6):721-9. doi: 10.1016/j.semarthrit.2013.11.003. Epub 2013 Nov 13. PMID 24332117